CLINICAL TRIAL: NCT06369142
Title: Intracoronary Stenting and Additional Results Achieved by ShockWAVE Coronary Lithotripsy: A Randomized, Multicenter Study About the Additional Benefit of Coronary Lithotripsy
Brief Title: Intracoronary Stenting and Additional Results Achieved by ShockWAVE Coronary Lithotripsy
Acronym: ISAR-WAVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Gemeinsamer Bundesaussschuss (Unknown); EvidentIQ Germany GmbH (Unknown); Monitoring Services GmbH (Unknown); Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GE IDE No. L00123
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Calcified lesion; Percutaneous Coronary Intervention; Stent; Intravascular Lithotripsy
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study participant as well as the follow-up physicians and site personal are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lesion preparation using coronary intravascular lithotripsy (Experimental)
  Interventions: Device: Intravascular lithotripsy (IVL)
- Lesion preparation using other methods than intravascular lithotripsy (Active Comparator): e.g. cutting or super high pressure balloons and/or ablative procedures
  Interventions: Device: Standard non-IVL methods

INTERVENTIONS:
Device: Intravascular lithotripsy (IVL) — Intravascular lithotripsy (IVL) and ballons with a nominal rated burst pressure of ≤ 18 atm
  Arms: Lesion preparation using coronary intravascular lithotripsy
Device: Standard non-IVL methods — Standard non-IVL methods treating severely calcified lesions such as special high, super high and cutting balloons and ablative procedures
  Arms: Lesion preparation using other methods than intravascular lithotripsy

SUMMARY:
The clinical trial is intended to evaluate the efficacy, safety and economic benefit of coronary lithotripsy compared to other additional procedures (cutting or super high pressure balloon angioplasty, ablative procedures) in lesion preparation and interventional treatment of severely calcified coronary stenoses.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥18 years and able to give informed consent
2. written informed consent to participate in the clinical trial
3. typical angina pectoris or non-invasive evidence of relevant ischemia under optimal drug therapy
4. angiographic evidence of coronary artery disease
5. de novo lesion in a native coronary artery
6. target vessel diameter 2.5-4 mm
7. severe calcification of the target lesion (angiographic grade 3)

Exclusion Criteria:

1. myocardial infarction <1 week
2. thrombus in the target vessel
3. life expectancy due to other disease <1 year
4. simultaneous participation in a clinical trial with medical devices or medicinal products that has not yet been completed
5. pregnancy (current, suspected, planned) or positive pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint of major cardiac and cerebrovascular events | 12 months after randomization
  all-cause mortality, non-fatal myocardial infarction, non-fatal stroke, clinically indicated revascularisation of the target vessel

SECONDARY OUTCOMES:
Mortality | 12 months after randomization
Cardiac mortality | 12 months after randomization
Non-fatal myocardial infarction | 12 months after randomization
Non-fatal stroke | 12 months after randomization
Clinically indicated target vessel revascularization | 12 months after randomization
Definite stent thrombosis | 12 months after randomization
Clinically indicated non-target vessel revascularization | 12 months after randomization
Hospitalization due to acute coronary syndrome | 12 months after randomization
Symptoms of coronary heart disease (CHD): physical health status | 12 months after randomization
Symptoms of CHD: mental health status | 12 months after randomization
Bleeding during index hospitalization or ≤30 days (BARC 3-5) | 30 days after randomization
Procedural failure (failed application of study-related additional procedure, final TIMI flow <3, >30% residual stenosis, vessel perforation, stent loss, stent delivery failure) | 12 months after randomization
Medical costs (index hospitalization and costs for re-hospitalization due to acute coronary syndrome) | 12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kastrati, MD, Study Chair — Deutsches Herzzentrum München, Klinik für Herz- und Kreislauferkrankungen
Locations (22):
- Germany (22):
  - Universitätsklinikum Heidelberg, Klinik für Kardiologie, Angiologie und Pneumologie, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Mannheim GmbH, I. Medizinische Klinik, Kardiologie, Angiologie, Hämostaseologie, Internistische Intensivmedizin, Mannheim, Baden-Wurttemberg
  - Hegau-Bodensee-Klinikum Singen GmbH, I. Medizinsche Klinik (Kardiologie und internistische Intensivmedizin), Singen, Baden-Wurttemberg
  - Cardiologikum Herzklinik Ulm MVZ, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Augsburg A.ö.R., Augsburg, Bavaria
  - Helios Amper-Klinikum Dachau, Kardiologie und Pneumologie, Dachau, Bavaria
  - Klinikum Landkreis Erding, Erding, Bavaria
  - Klinikum Ingolstadt, Ingolstadt, Bavaria
  - Deutsches Herzzentrum München, Munich, Bavaria
  - Klinikum der Ludwig-Maximilians-Universität München, München, Bavaria
  - Augustinum Klinik München, München, Bavaria
  - Krankenhaus Landshut-Achdorf, LAKUMED Kliniken, Landshut, Germany
  - Universitäres Herz- und Gefäßzentrum, Hamburg, Hamburg
  - Klinikum Hersfeld Rotenburg GmbH Herz-Kreislauf-Zentrum Institut für Klinische Forschung, Rotenburg an der Fulda, Hesse
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen, North Rhine-Westphalia
  - Elisabeth Krankenhaus Essen Contilia Herz- und Gefäßzentrum Klinik für Kardiologie und Angiologie Kardiovaskuläres Studienzentrum, Essen, North Rhine-Westphalia
  - Krankenhaus Barmherzige Brüder Trier, Trier, Rhineland-Palatinate
  - Herzzentrum Dresden GmbH Universitätsklinik an der Technischen Universität Dresden, Dresden, Saxony
  - Asklepios Klinik Bad Oldesloe Innere Medizin, Kardiologie und Intensivmedizin, Bad Oldesloe, Schleswig-Holstein
  - Klinik für Kardiologie, Angiologie und Intensivmedizin Deutsches Herzzentrum der Charité, Berlin, State of Berlin
  - BG Klinikum Unfallkrankenhaus Berlin gGmbH, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cassese S, Simonetti F, Covarrubias HAA, Janisch M, Joner M, Kufner S, Lenz T, Pellegrini C, Rheude T, Sager H, Schunkert H, Starnecker F, Voll F, Xhepa E, Kastrati A, Kessler T. Intracoronary stenting and additional results achieved by shockWAVE coronary lithotripsy: design and rationale of ISAR-WAVE trial. Am Heart J. 2025 Apr;282:1-12. doi: 10.1016/j.ahj.2024.12.008. Epub 2024 Dec 20. PMID 39710352